CLINICAL TRIAL: NCT07176117
Title: Surfactant Prophylaxis in LAte Preterm to Early Term Infants Using a Supraglottic Airway Device to Help Improve Outcomes
Brief Title: Surfactant Using a Supraglottic Airway Device in Late Preterm to Early Term Infants
Acronym: SPLASH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Principal Investigator, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPLASH
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Syndrome (Neonatal); Surfactant
Keywords: supraglottic airway device
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prophylactic Surfactant (Experimental): A single dose of surfactant (Curosurf) will be given via Surfactant Administration Through Laryngeal or Supraglottic Airways (SALSA). Infants who receive SALSA will remain on non-invasive respiratory support (Continuous Positive Airway Pressure).
  Interventions: Procedure: Surfactant Administration Through Laryngeal or Supraglottic Airway (SALSA)
- Expectant Management (CPAP) (Active Comparator): For participating infants randomly assigned to receive continuation of non-invasive respiratory support, they will remain on continuous positive airway pressure (CPAP).
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Procedure: Surfactant Administration Through Laryngeal or Supraglottic Airway (SALSA) — A single dose of surfactant will be given via Surfactant Administration Through Laryngeal or Supraglottic Airways (SALSA). A supraglottic airway device will be used as a standardized procedure for surfactant administration via SALSA using an AirLife Air-Q.
  Arms: Prophylactic Surfactant
Procedure: Continuous Positive Airway Pressure (CPAP) — Infants to receive continuation of non-invasive respiratory support will remain on continuous positive airway pressure (CPAP).
  Arms: Expectant Management (CPAP)

SUMMARY:
The purpose of this research is to learn new information that may help other infants that have respiratory distress syndrome and need breathing support after birth. The goal of this research is to see if continuous positive airway pressure (CPAP) alone or CPAP with surfactant administration through a less invasive method via an Airway Device (supraglottic airway device) temporarily placed above the vocal cords is better for treating respiratory distress syndrome in late preterm and early term infants.

ELIGIBILITY:
Inclusion Criteria:

* Newborns 33-38+6 weeks gestation at birth
* ≤ 6 hours old
* Respiratory Distress: [Silverman Andersen Score (SAS) ≥ 5, or Respiratory Severity Score (RSS) ≥ 1.25]
* Clinical decision for non-invasive respiratory support
* Written parental consent

Exclusion Criteria:

* Surrogate deliveries
* Major congenital or chromosomal anomalies
* Prior intubation or receipt of surfactant
* Known or suspected hypoxic ischemic encephalopathy (HIE)
* Known or suspected neuromuscular disorder
* Unanticipated survival

Ages: 33 Weeks to 38 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 422 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Ranked Composite of Morbidities | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Determine if there is a difference in ranked composite of morbidities including death, development of pneumothorax/ pulmonary air leaks, Respiratory Severity Score (RSS), time to initial feeding, and LOS (length of hospital stay) between the treatment and control groups using a linked count of participants who fall within each prespecified rank.

SECONDARY OUTCOMES:
Length of Hospital Stay | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Length of hospital stay (LOS), days.

OTHER OUTCOMES:
Time to Parent Bonding | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Time to parent bonding from initial parent skin-to-skin contact.
Duration of Mechanical Ventilation | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Total duration of mechanical ventilation (MV) with endotracheal tube, days.
Duration of Continuous Positive Airway Pressure | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Total duration of Continuous Positive Airway Pressure (CPAP), days.
Duration of Non-Invasive Respiratory Support | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Duration of non-invasive respiratory support with positive pressure and/or high flow, days.
Oxygen Administration | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Oxygen administration requirements for Fraction of Inspired Oxygen (FiO2).
CPAP Failure | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  CPAP (Continuous Positive Airway Pressure) Failure, defined using any of the following: Respiratory Severity Score (RSS), Silverman Andersen (SAS), Respiratory acidosis, or Severe apnea.
Surfactant Administration | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Surfactant administration (additional dose administered to infants randomized to receive surfactant or any surfactant to infants receiving expectant CPAP management).
Time to Initial Feed | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Time to initial breastfeeding (including dry or nutritive) or oral feeding.
Time to Full Feeds | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Time to full feeds i.e. no parenteral nutrition.
Incidence of Pneumothorax | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Incidence of pneumothorax/ pulmonary air leaks.
Incidence of Late Onset Sepsis | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Incidence of late onset sepsis.
Maternal Length of Stay | From hospital admission to study completion at hospital discharge after birth.
  Maternal total length of stay.
Feeds at discharge | From date of birth (day of life 1) through study completion at birth-hospital discharge, up to 6 months of age.
  Breastfeeding at time of discharge (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (3):
- United States (3):
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, particularly data that underlie the results reported in this article after deidentification will be available with other researchers, including data dictionaries for meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Data and publication are available at http://clinicaltrials.gov
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Ho JJ, Subramaniam P, Davis PG. Continuous positive airway pressure (CPAP) for respiratory distress in preterm infants. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD002271. doi: 10.1002/14651858.CD002271.pub3. PMID 33058208
- [Background] Polin RA, Carlo WA; Committee on Fetus and Newborn; American Academy of Pediatrics. Surfactant replacement therapy for preterm and term neonates with respiratory distress. Pediatrics. 2014 Jan;133(1):156-63. doi: 10.1542/peds.2013-3443. Epub 2013 Dec 30. PMID 24379227
- [Background] Dargaville PA, Kamlin COF, Orsini F, Wang X, De Paoli AG, Kanmaz Kutman HG, Cetinkaya M, Kornhauser-Cerar L, Derrick M, Ozkan H, Hulzebos CV, Schmolzer GM, Aiyappan A, Lemyre B, Kuo S, Rajadurai VS, O'Shea J, Biniwale M, Ramanathan R, Kushnir A, Bader D, Thomas MR, Chakraborty M, Buksh MJ, Bhatia R, Sullivan CL, Shinwell ES, Dyson A, Barker DP, Kugelman A, Donovan TJ, Tauscher MK, Murthy V, Ali SKM, Yossuck P, Clark HW, Soll RF, Carlin JB, Davis PG; OPTIMIST-A Trial Investigators. Effect of Minimally Invasive Surfactant Therapy vs Sham Treatment on Death or Bronchopulmonary Dysplasia in Preterm Infants With Respiratory Distress Syndrome: The OPTIMIST-A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2478-2487. doi: 10.1001/jama.2021.21892. PMID 34902013
- [Background] Ramaswamy VV, Bandyopadhyay T, Abiramalatha T, Pullattayil S AK, Szczapa T, Wright CJ, Roehr CC. Clinical decision thresholds for surfactant administration in preterm infants: a systematic review and network meta-analysis. EClinicalMedicine. 2023 Jul 20;62:102097. doi: 10.1016/j.eclinm.2023.102097. eCollection 2023 Aug. PMID 37538537
- [Background] Ramaswamy VV, Abiramalatha T, Bandyopadhyay T, Boyle E, Roehr CC. Surfactant therapy in late preterm and term neonates with respiratory distress syndrome: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2022 Jul;107(4):393-397. doi: 10.1136/archdischild-2021-322890. Epub 2021 Oct 22. PMID 34686533
- [Background] Calevo MG, Veronese N, Cavallin F, Paola C, Micaglio M, Trevisanuto D. Supraglottic airway devices for surfactant treatment: systematic review and meta-analysis. J Perinatol. 2019 Feb;39(2):173-183. doi: 10.1038/s41372-018-0281-x. Epub 2018 Dec 5. PMID 30518796
- [Background] Lockyear C, Coe K, Greenberg RG, Clark RH, Aleem S. Trends in morbidities of late preterm infants in the neonatal intensive care unit. J Perinatol. 2023 Nov;43(11):1379-1384. doi: 10.1038/s41372-023-01705-5. Epub 2023 Jul 1. PMID 37393396
- [Background] Katheria A, Ines F, Banerji A, Hopper A, Uy C, Chundu A, Coughlin K, Hutson S, Morales A, Sauberan J, Poeltler D, Dorner R, Rich W, Finer N. Caffeine and Less Invasive Surfactant Administration for Respiratory Distress Syndrome of the Newborn. NEJM Evid. 2023 Dec;2(12):EVIDoa2300183. doi: 10.1056/EVIDoa2300183. Epub 2023 Nov 21. PMID 38320499
- [Background] Jackson W, Taylor G, Bamat NA, Zimmerman K, Clark R, Benjamin DK, Laughon MM, Greenberg RG, Hornik CP. Outcomes associated with surfactant in more mature and larger premature infants with respiratory distress syndrome. J Perinatol. 2020 Aug;40(8):1171-1177. doi: 10.1038/s41372-020-0625-1. Epub 2020 Feb 20. PMID 32080333
- [Background] Berger DS, Garg B, Penfield CA, Caughey AB. Respiratory distress syndrome is associated with increased morbidity and mortality in late preterm births. Am J Obstet Gynecol MFM. 2024 Jun;6(6):101374. doi: 10.1016/j.ajogmf.2024.101374. Epub 2024 Apr 5. PMID 38583712
- [Background] Olivier F, Nadeau S, Caouette G, Piedboeuf B. Association between Apnea of Prematurity and Respiratory Distress Syndrome in Late Preterm Infants: An Observational Study. Front Pediatr. 2016 Sep 26;4:105. doi: 10.3389/fped.2016.00105. eCollection 2016. PMID 27725928
- [Background] Consortium on Safe Labor; Hibbard JU, Wilkins I, Sun L, Gregory K, Haberman S, Hoffman M, Kominiarek MA, Reddy U, Bailit J, Branch DW, Burkman R, Gonzalez Quintero VH, Hatjis CG, Landy H, Ramirez M, VanVeldhuisen P, Troendle J, Zhang J. Respiratory morbidity in late preterm births. JAMA. 2010 Jul 28;304(4):419-25. doi: 10.1001/jama.2010.1015. PMID 20664042
- [Background] Spong CY, Mercer BM, D'Alton M, Kilpatrick S, Blackwell S, Saade G. Timing of indicated late-preterm and early-term birth. Obstet Gynecol. 2011 Aug;118(2 Pt 1):323-333. doi: 10.1097/AOG.0b013e3182255999. PMID 21775849